CLINICAL TRIAL: NCT05671159
Title: COMPArative Study of the Consequence on innaTe Immune Response du to Bacterial or Viral Infection in Patients Admitted to Intensive Care Unit
Acronym: COMPACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 87RI22_0031(COMPACT)
Record Dates: First submitted 2022-10-28; First posted 2023-01-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Viral Infection; Sepsis
Keywords: bacteria; virus; Immune response; acute infection; immature granulocyte
MeSH Terms: conditions — Virus Diseases; Sepsis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bacterial infection (Experimental)
  Interventions: Other: Blood sample
- viral infection (Other)
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — A supplementary blood sample will be taken including a 5mL EDTA tube and a paxgene tube

SUMMARY:
Patient admitted in intensive care unit (ICU) for acute infection whether it be viral or bacterial had major impairment of the immune response. One hallmark of the immune impairment is presence of immature granulocyte (IG) in blood. Depend of initial trigger (virus or bacteria) concentration, phenotype and function of IG seems to be different. In this prospective trial, immature granulocytes will be analyzed in depth in immunocompetent patients hospitalized in the intensive care unit for an acute viral or bacterial infection.

DETAILED DESCRIPTION:
Granulocytes are a key actor of immune response during acute viral or bacterial infection. During their maturation in bone marrow they went from immature form to mature form. In physiological condition only mature form are present in blood. However, in case of acute viral or bacterial infection, immature granulocytes (CD10low/CD16low) could be released in blood. But concentration, phenotype and function of these IG seems to be different between bacterial and viral infection. Indeed, in bacterial infection, concentration of IG is high (> 20%) and they expressed CD64 and CD123. In case of viral infection, blood concentration of IG is lower and they expressed CD62-L. These phenotype differences are probably associated with functional modification. A more precise characterization of the phenotype and functions of IG according to the stimulus (bacterial or viral) could provide a better understanding of the innate immune response in patients hospitalized in ICU for acute infection. The investigators will analysis by flow cytometry IG subsets (PDL1 CD62L LOX-1 CD45 CD64 CD15 CD123 CD16 CD10 CRTH2) of adult immunocompetent patient hospitalized in ICU for less than 24 hours for acute infection. Transcriptomic and cytokine analysis will be also performed. Infectious status will be validated by a blind adjudication committee which will classify patient in certain bacterial infection, certain viral infection, co-infection and no confirmed infection.

ELIGIBILITY:
Inclusion Criteria:

* Bacterial infection:

  * Adult patient hospitalized for less than 24 hours in ICU for community documented sepsis
  * Vasopressor support
  * SOFA score > 4
* Viral infection:

  * Adult patient hospitalized for less than 24 hours in ICU for confirmed viral acute infection.
  * High flow oxygen, non-invasive or invasive ventilation since less than 24 hours
  * Moderate to severe ARDS with PaO2/FiO2 < 200mmHg and a FiO2 ≥ 0.6.

Exclusion Criteria:

* Bacterial infection:

  * Antibiotics or hospitalized in ICU in the previous 3 months
  * Immunocompromized patient
  * Ongoing acute or chronic viral infection
* Viral infection:

  * Antibiotics or hospitalized in ICU in the previous 3 months
  * Immunocompromized patient
  * Current antibiotics
  * Ongoing chronic viral infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-02-19 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Granules expressing CD123 and CD64 | Day 0
  Measurement by flow cytometry of the percentage of granules expressing CD123 and CD64 depending on the type of infection (viral or bacterial).

SECONDARY OUTCOMES:
granules expressing CD62-L | Day 0
  Measurement by flow cytometry of the percentage of granules expressing CD62-L according to the type of infection (viral or bacterial).
Immune functions genes expression | Day 0
  Evaluate the expression of genes related to immune functions of the different subpopulations of immature granules by measuring the amount of mRNA
blood concentrations of cytokines | Day 0
  Measurement by multiplex Elisa-test of blood cytokine concentrations (IL-8, IL-1, IL-12p70, IL-6, IL-10, IP-10, TNF-a, IFN-g)
blood concentrations of activation markers | Day 0
  Measurement by multiplex Elisa test of blood concentrations of activation markers (RETN, LCN2, HGF; G-CSF)
Sequential Organ Failure Assessment (SOFA) score | Day 0
  Evolution of a modified Sequential (Sepsis-Related) Organ Failure Assessment (SOFA) score (no gradation of the neurologic system) at day 0. Min value =0. Max value =20 . The highest score means the worst situation

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges University Hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No